CLINICAL TRIAL: NCT00075270
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, 2-Arm, Phase III Study of Oral GW572016 in Combination With Paclitaxel in Subjects Previously Untreated or Advanced or Metastatic Breast Cancer
Brief Title: Paclitaxel With / Without GW572016 (Lapatinib) As First Line Therapy For Women With Advanced Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGF30001; NCT00085046 (obsolete NCT alias)
Record Dates: First submitted 2004-01-07; First posted 2004-01-09 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms, Breast
Keywords: metastatic breast cancer; ErbB1; kinase inhibitor; ErbB2; EGFR; lapatinib; Her2-neu
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Lapatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Lapatinib 1500 mg, once daily and Paclitaxel 175 mg/m Intravenously over 3 hours ever 3 weeks
  Interventions: Drug: Paclitaxel; Drug: GW572016 (Lapatinib)
- Arm 2 (Placebo Comparator): Paclitaxel 175 mg/m Intravenously over 3 hours ever 3 weeks and Placebo
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Active Comparator
Drug: GW572016 (Lapatinib) — Oral GW572016 Lapatinib
  Other Names: Paclitaxel
  Arms: Arm 1

SUMMARY:
The purpose of this study is to determine the efficacy and safety of an oral dual tyrosine kinase inhibitor (GW572016) in combination with paclitaxel compared to paclitaxel alone in first line advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Signed Informed Consent
* Able to swallow an oral medication
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram
* Adequate kidney and liver function
* Adequate bone marrow function
* Tumor tissue available for testing
* Prior adjuvant or neoadjuvant therapy is permitted with an anthracycline or anthracenedione-containing regimen however, subjects must have had cumulative doses of less than 360 mg/m2 of doxorubicin, 720 mg/m2 of epirubicin, or 72 mg/m2 of mitoxantrone
* No Her2/neu overexpression in tumor tissue tested or status unknown if tissue has never been tested

Exclusion criteria:

* Prior treatment regimens for advanced or metastatic breast cancer.
* Pregnant or lactating
* Conditions that would effect the absorption of an oral drug
* Active infection
* Brain metastases
* Treatment with EGFR (Endothelial Growth Factor Receptor) inhibitor.
* Known hypersensitivity to Taxol or excipients of Taxol
* Peripheral neuropathy of Grade 2 or greater is not permitted
* Severe Cardiovascular disease or cardiac disease requiring a device.
* Serious medical or psychiatric disorder that would interfere with the patient's safety or informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2004-01; Primary Completion 2006-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (152):
- United States (43):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Port Saint Lucie, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Nyack, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
- Australia (4):
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Wodonga, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- GSK Investigational Site, Vienna, Austria
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Brazil (2):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
- Canada (5):
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
- Germany (17):
  - GSK Investigational Site, Aalen, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Coburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Fürstenwalde, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Stade, Lower Saxony
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Ibbenbueren, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Jena, Thuringia
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Zalaegerszeg-Pózva
- Italy (15):
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Forlì, Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Pietra Ligure (SV), Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Candiolo (TO), Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Prato (PO), Tuscany
  - GSK Investigational Site, Perugia, Umbria
- Latvia (3):
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
- Mexico (4):
  - GSK Investigational Site, Colima, Colima
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Acapulco de Juárez, Guerrero
  - GSK Investigational Site, Guadalajara, Jalisco
- Netherlands (4):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Utrecht
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
- GSK Investigational Site, Lahore, Pakistan
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao
- Poland (5):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Moscow Region
  - GSK Investigational Site, Saint Petersburg
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Poprad
- South Africa (5):
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Capital Park
  - GSK Investigational Site, Overport
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Port Elizabeth
- South Korea (2):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (14):
  - GSK Investigational Site, Alcorcón/Madrid
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Cuidad Real
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Las Palmas de Gran Canaria
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Zaragoza
- GSK Investigational Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Tenori L, Oakman C, Claudino WM, Bernini P, Cappadona S, Nepi S, Biganzoli L, Arbushites MC, Luchinat C, Bertini I, Di Leo A. Exploration of serum metabolomic profiles and outcomes in women with metastatic breast cancer: a pilot study. Mol Oncol. 2012 Aug;6(4):437-44. doi: 10.1016/j.molonc.2012.05.003. Epub 2012 Jun 1. PMID 22687601
- [Background] Finn RS, Press MF, Dering J, Arbushites M, Koehler M, Oliva C, Williams LS, Di Leo A. Estrogen receptor, progesterone receptor, human epidermal growth factor receptor 2 (HER2), and epidermal growth factor receptor expression and benefit from lapatinib in a randomized trial of paclitaxel with lapatinib or placebo as first-line treatment in HER2-negative or unknown metastatic breast cancer. J Clin Oncol. 2009 Aug 20;27(24):3908-15. doi: 10.1200/JCO.2008.18.1925. Epub 2009 Jul 20. PMID 19620495
- [Derived] Sherrill B, Di Leo A, Amonkar MM, Wu Y, Zvirbule Z, Aziz Z, Bines J, Gomez HL. Quality-of-life and quality-adjusted survival (Q-TWiST) in patients receiving lapatinib in combination with paclitaxel as first-line treatment for metastatic breast cancer. Curr Med Res Opin. 2010 Apr;26(4):767-75. doi: 10.1185/03007991003590860. PMID 20095796

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 580 participants were enrolled and randomized to treatment; however one participant withdrew from the study before taking any medication. Thus, only 579 participants were included in the Intent-to-Treat Population (comprised of all randomized participants who had received at least one dose of randomized therapy [lapatinib or placebo]).
Groups:
- Lapatinib With Paclitaxel: Participants received lapatinib 1500 milligrams (mg) orally once daily (OD) with paclitaxel 175 mg/meters squared (m^2) intravenously (IV) over the course of 3 hours, every 3 weeks. The treatment group was stratified by sites of metastatic disease and stage of disease. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
- Placebo With Paclitaxel: Participants received matching placebo orally OD with paclitaxel (175 mg/m^2 IV) over the course of 3 hours, every 3 weeks. The treatment group was stratified by sites of metastatic disease and stage of disease. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
Period: Overall Study
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Started | 291 | 288
Missing | 26 (These participants have no completion status information recorded on the case report forms.) | 13 (These participants have no completion status information recorded on the case report forms.)
Completed | 5 | 4
Not Completed | 286 | 284
Not completed — Withdrawal by Subject | 28 | 21
Not completed — Lost to Follow-up | 25 | 28
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 198 | 215
Not completed — Other/Unknown | 9 | 5
Not completed — Missing | 26 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel | Total
Number analyzed (Participants) | 291 | 288 | 579
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (10.45) | 52.4 (10.98) | 51.8 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 288 | 579
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 190 | 182 | 372
  Black | 10 | 10 | 20
  Asian | 30 | 35 | 65
  American Hispanic | 54 | 53 | 107
  Unknown | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression as Evaluated by the Investigator
Description: Time to progression (TTP) is defined as the interval between the date of randomization and the earliest date of progression of disease (PD) or death due to breast cancer. The investigator assessed PD based on radiological PD (imaging data) and clinical symptomatic progress (Response Evaluation Criteria in Solid Tumors [RECIST] Criteria: target lesion (TL), at least a 20% increase in the sum of largest diameter (LD) of TLs or the appearance of one or more new lesions; non-TL (NTL), the appearance of one or more new lesions and/or unequivocal progression of existing NTLs). TTP was assessed in participants who died due to breast cancer or progressed, as assessed by the investigator, as well as in those who were censored and completed follow-up and those who were censored but are still being followed. For censored participants (those without a documented date of disease progression/death due to breast cancer), the date of the last radiographic assessment was used.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: Intent-to-Treat (ITT) Population: all randomized participants who had received at least one dose of randomized therapy (lapatinib or placebo)
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
weeks | 29.0 [13.9 to 46.9] | 22.9 [12.0 to 38.3]
Statistical Analysis 1: Comparison: Lapatinib With Paclitaxel vs Placebo With Paclitaxel; Test type: Superiority or Other; p = 0.142, Log Rank — P-value from stratified log-rank test, stratifying for stage of disease and site of disease at screening; Hazard Ratio, log = 0.87, 95% CI 2-sided [0.72 to 1.05] — The estimate of the treatment hazard ratio is based on the log-rank test

2. Primary Outcome: Time to Progression as Evaluated by the Independent Review Committee (IRC)
Description: Time to progression is defined as the interval between the date of randomization and the earliest date of progression of disease (PD) or death due to breast cancer. The IRC assessed PD based on radiological PD (imaging data) and clinical symptomatic progress (Response Evaluation Criteria in Solid Tumors [RECIST] Criteria: target lesion (TL), at least a 20% increase in the sum of largest diameter (LD) of TLs or the appearance of one or more new lesions; non-TL (NTL), the appearance of one or more new lesions and/or unequivocal progression of existing NTLs). TTP was assessed in participants who died due to breast cancer or progressed, as assessed by the independent reviewer, as well as in those who were censored and completed follow-up and those who were censored but are still being followed. For censored participants (those without a documented date of disease progression/death due to breast cancer), the date of the last radiographic assessment was used.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Lapatinib With Paclitaxel: Participants received lapatinib 1500 mg orally OD with paclitaxel 175 m^2 IV over the course of 3 hours, every 3 weeks. The treatment group was stratified by sites of metastatic disease and stage of disease. Participants were treated until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
weeks | 33.7 [18.7 to 69.1] | 26.1 [12.9 to 57.1]
Statistical Analysis 1: Comparison: Lapatinib With Paclitaxel vs Placebo With Paclitaxel; Test type: Superiority or Other; p = 0.094, Log Rank — P-value from stratified log-rank test, stratifying for stage of disease and site of disease at screening; Hazard Ratio, log = 0.82, 95% CI 2-sided [0.65 to 1.04] — The estimate of the treatment hazard ratio was based on the log-rank test

3. Secondary Outcome: Number of Participants With Tumor Response as Evaluated by the Investigator
Description: The percentage of participants with tumor response is defined as those participants with measurable disease who achieved either a complete response (CR) or partial response (PR). The Response Evaluation Criteria in Solid Tumors (RECIST) was used to evaluate the measurability of tumor lesions, to determine target lesion (TLs) and non-target lesion (NTLs). CR (TLs and NTLs): the disappearance of all TLs and NTLs; PR (for TLs): at least a 30% decrease in the sum of the largest diameter (LD) of TLs, taking as a reference the Baseline sum LD; PR (for NTLs): persistence of one or more lesions.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  CR | 14 | 6
  PR | 88 | 67

4. Secondary Outcome: Number of Participants With Tumor Response as Evaluated by the Independent Review Committee
Description: The percentage of participants with tumor response is defined as those participants with measurable disease who achieved either a complete response (CR) or partial response (PR). The RECIST criteria was used to evaluate the measurability of tumor lesions, to determine target lesion (TLs) and non-target lesion (NTLs). CR (TLs and NTLs): the disappearance of all TLs and NTLs; PR (for TLs): at least a 30% decrease in the sum of the largest diameter (LD) of TLs, taking as a reference the Baseline sum LD; PR (for NTLs): persistence of one or more lesions.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  CR | 1 | 1
  PR | 77 | 53

5. Secondary Outcome: Percentage of Participants With Clinical Benefit (CB) as Assessed by the Investigator
Description: Percentage of participants. with CB is defined as the percentage of participants with evidence of CR (disappearance of all TLs and NTLs), PR (TLs: a >=30% decrease in the sum of the LD, taking as a reference the Baseline sum LD; NTLs: persistence of >=1 lesion), or stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) for >=6 months based on RECIST criteria. PD for TL: a >=20% increase in the sum of the LD of TLs or the appearance of >=1 new lesion. PD for NTLs: the appearance of >=1 new lesion and/or unequivocal progression of existing NTLs.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
Percentage of participants | 40.5 | 31.9

6. Secondary Outcome: Number of Participants With a Response of CR or PR by the Indicated Study Week
Description: Time to response (TTR) is defined as the time from randomization until the first documented evidence of CR (disappearance of all TLs and NTLs) or PR (for TLs: a >=30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD; for NTLs: the persistence of >=1 lesion) (whichever status was recorded first). TTR data are displayed as the number of participants achieving a CR or PR by the indicated week. The investigator evaluated the TTR, and the analysis was based on responses confirmed at a repeat assessment, with the TTR taken as the first time the response was observed.
Time Frame: Weeks 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, and 72
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  Week 6 | 3 | 0
  Week 12 | 83 | 55
  Week 18 | 86 | 57
  Week 24 | 98 | 69
  Week 30 | 98 | 69
  Week 36 | 101 | 71
  Week 42 | 102 | 72
  Week 48 | 102 | 72
  Week 54 | 102 | 72
  Week 60 | 102 | 72
  Week 66 | 102 | 72
  Week 72 | 102 | 73

7. Secondary Outcome: Duration of Response (DOR)
Description: The investigator evaluated the DOR for the subset of participants who showed a CR (disappearance of all TLs and NTLs) or PR (TLs: a >=30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD; NTLs: persistence of >=1 lesion). DOR is defined as the time from the first documented evidence of PR or CR until the first documented sign of PD (TL: a >=20% increase in the sum of the LD of TLs or the appearance of >=1 new lesion; NTL: the appearance of >=1 new lesion and/or unequivocal progression of existing NTLs) or death due to breast cancer, if sooner.
Time Frame: From the time of the first documented complete or partial response until the first documented evidence of progression or death (average of 26 weeks)
Population: ITT Population. Only participants who had a CR or PR were evaluated.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 102 | 73
weeks | 28.3 [22.3 to 50.0] | 27.1 [18.1 to 46.3]

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the interval between the date of randomization and the earliest date of progression disease (PD) or death due to any cause, if sooner. For TLs, progressive disease is defined as at least a 20% increase in the sum of the LD of TLs or the appearance of 1 or more new lesions. For NTLs, progressive disease is defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. par., participants.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population. PFS was assessed in par. who died or progressed, as well as in those who were censored and completed follow-up and those who were censored but are still being followed. For censored par. (those without a documented date of disease progression/death due to any cause), the date of the last radiographic assessment was used.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
weeks | 25.1 [21.9 to 32.1] | 22.6 [21.0 to 25.4]

9. Secondary Outcome: Number of Participants Who Progressed or Died at or Prior to 6 Months, as a Measure of Six Months Progression-free Survival (PFS)
Description: PFS is defined as the interval between the date of randomization and the earliest date of disease progression or death due to any cause, if sooner. Six months PFS is defined as PFS at six months from the time of randomization. Raw data for 6 months PFS are not available; thus, data are presented as the number of participants who progressed or died at or prior to 6 months. For TLs, progressive disease is defined asat least a 20% increase in the sum of the LD of TLs or the appearance of 1 or more new lesions. For NTLs, progressive disease is defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. PFS was assessed in participants who died or progressed, as well as in those who were censored and completed follow-up and those who were censored but are still being followed. For censored participants (those without a documented date of disease progression/death due to breast cancer), the date of the last radiographic assessment was used.
Time Frame: Randomization until the date of disease progression or death (average of 26 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants | 133 | 153

10. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: Randomization until the date of death due to any cause (average of 24 months)
Population: ITT population. Overall survival was assessed in participants who died as well as in those who were censored and completed follow-up and those who were censored but are still being followed. For censored participants (those still alive), the date of the last contact was used.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
months | 23.82 [19.88 to 26.18] | 20.17 [17.84 to 23.92]

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) Questionnaire Scores
Description: The FACT-B questionnaire was designed to measure multidimensional quality of life (QOL) in participants with breast cancer. The physical and functional well-being subscale scores range from 0 to 28, based on 7 questions (each scored from 0 [not at all] to 4 [very much] for all subscales); the emotional and social/family well-being (1 question optional) subscale scores range from 0 to 24 (based on 6 questions), and the additional concerns subscale score ranges from 0 to 40, based on 10 questions. The FACT-B Total Score (0 [better QOL] to 144 [worse QOL]) is the sum of the subscale scores.
Time Frame: Baseline (Day 1); Weeks 9, 21, 33, and 45; Withdrawal
Population: ITT Population. Only participants contributing data at the indicated time points were analyzed. Only observed data were collected, and score analyses were conducted using the last observation carried forward (LOCF) method: the last available on-therapy observation for a participant was used to estimate missing data points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 208 | 230
Scores on a scale
  Week 9, n=208, 230 | -1.1 (16.09) | -2.3 (16.27)
  Week 21, n=126, 125 | 1.0 (16.63) | -1.3 (17.13)
  Week 33, n=72, 64 | 1.4 (17.39) | -2.0 (12.75)
  Week 45, n=35, 38 | 2.3 (22.05) | -1.4 (10.79)
  Withdrawal, n=190, 212 | -5.0 (19.53) | -8.4 (17.99)

12. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire Scores
Description: The FACT-G questionnaire was designed to measure multidimensional QOL in participants with cancer and includes subscales for physical, social/family, emotional, and functional well-being. The physical, social/family, and functional well-being subscale scores range from 0 to 28, based on responses to 7 questions (each question scored from 0 [not at all] to 4 [very much]); the emotional well-being subscale score ranges from 0 to 24, based on responses to 6 questions. The FACT-G Total Score (ranging from 0 [better QOL] to 108 [worse QOL]) is the sum of the subscale scores.
Time Frame: Baseline (Day 1); Weeks 9, 21, 33, and 45; Withdrawal
Population: ITT Population. Only participants contributing data at the indicated time points were analyzed. Only observed data were collected, and score analyses were conducted using the LOCF method.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 213 | 232
Scores on a scale
  Week 9, n=213, 232 | -0.7 (13.35) | -1.3 (13.26)
  Week 21, n=127, 125 | 0.4 (13.97) | -0.2 (14.38)
  Week 33, n=71, 65 | 1.1 (14.80) | -1.7 (10.81)
  Week 45, n=34, 39 | 0.9 (17.68) | -1.6 (10.41)
  Withdrawal, n=193, 214 | -4.4 (16.11) | -7.5 (15.02)

13. Secondary Outcome: Change From Baseline in Trial Outcome Index (TOI) Questionnaire Scores
Description: The TOI questionnaire was designed to measure multidimensional QOL in participants with cancer and includes subscales for physical, functional well-being, and additional cancer concerns. The physical and functional well-being subscale scores range from 0 to 28, based on 7 questions (each question scored from 0 [not at all] to 4 [very much]); the breast cancer unweighted subscale scores range from 0 to 36, based on 9 questions. The total TOI score (ranging from 0 [better QOL] to 92 [worse QOL]) is the sum of the TOI subscale scores.
Time Frame: Baseline (Day 1); Weeks 9, 21, 33, and 45; Withdrawal
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 208 | 232
Scores on a scale
  Week 9, n=208, 232 | -2.3 (12.32) | -2.6 (11.88)
  Week 21, n=126, 125 | -0.5 (11.99) | -2.7 (12.42)
  Week 33, n=72, 65 | -0.1 (12.83) | -2.9 (9.05)
  Week 45, n=36, 38 | 1.5 (15.91) | -2.8 (8.98)
  Withdrawal, n=190, 212 | -4.4 (14.30) | -6.1 (12.84)

14. Secondary Outcome: Number of Participants With the Indicated ErbB2 Status at Baseline
Description: The Press Laboratory collected tumor tissues of participants for ErbB2 testing. ErbB2 testing is done to detect breast cancer and predict its likely outcome. All samples were analyzed by the Press Laboratory. Participants were categorized as ErbB2 positive (overexpression of the ErbB2 gene), ErbB2 negative, and assay not done (which included participants with no available samples and those with inconclusive results). ErbB2 status is determined by immunohistochemistry (ICH) assay and fluorescence in situ hybridization (FISH) testing. Negative ErbB2 status is defined as 0 or 1+ by IHC, or as 2+ by IHC and FISH.
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  Positive | 52 | 39
  Negative | 199 | 202
  Assay not done | 40 | 47

15. Secondary Outcome: ErbB2 Ratio
Description: The Press Laboratory collected tumor tissues of participants for biomarker testing. All samples were analyzed by the Press Laboratory. The ratio of ErbB2 gene signals to chromosome 17 signals, which indicates the progression of breast cancer, was calculated. Low levels of amplification (few copies) may have a ratio of 2-5, whereas high levels of amplification may have a ratio >10.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio of signals
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 220 | 200
ratio of signals | 2.23 (2.301) | 2.14 (2.214)

16. Secondary Outcome: Number of Participants With the Indicated Immunohistochemistry (IHC) Results at Screening
Description: The Press Laboratory tested tumor tissue samples (taken at Screening, prior to randomization to study treatment) to determine intra-tumoral expression levels of ErbB1, ErbB2, and other analytes associated with these pathways by IHC, the process of detecting antigens (e.g., proteins) in cells of a tissue section. The IHC assessment is expressed as: 0, no staining (no cancer cells); 1+, faint staining; 2+, weak to moderate complete staining; 3+, strong complete staining (many cancer cells). A status of "Assay not done" was assigned to participants with no available samples and to those with inconclusive results. If strong staining is observed, breast cancer that has high levels of HER2 expression (overexpression) is indicated. If moderate/weak staining is observed (IHC=2+), breast cancer that has low/moderate expression levels is indicated. When no staining is observed (IHC=0), breast cancer HER2 expression may be below the level of detection of the assay.
Time Frame: Screening (Day -1)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  0 | 139 | 139
  1+ | 50 | 51
  2+ | 15 | 22
  3+ | 40 | 28
  Assay not done | 47 | 48

17. Secondary Outcome: Number of Participants With the Indicated ErbB2 Fluorescence in Situ Hybridization (FISH) Results
Description: The Press Laboratory tested participants who were 2+ (weak to moderate complete staining) or 3+ (strong complete staining) for ErbB2 overexpression by IHC for ErbB2 gene amplification using the FISH assay. The results of the FISH assay can be ErbB2 gene "amplification" (increased number of copies of the ErbB2 gene) or "non-amplification" (not many copies of the ErbB2 gene). A status of "Assay not done" was assigned to those participants with no available samples and to those with inconclusive results (e.g., due to hybridization or staining problems).
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 291 | 288
participants
  Amplified | 45 | 35
  Non-amplified | 175 | 165
  Assay not done | 71 | 88

18. Secondary Outcome: Serum ErbB1 Concentration
Description: The Quest Laboratory collected blood samples for quantitative determination of serum ErbB1. The results of serum monitoring were used to compare tumor response rates following randomized therapy.
Time Frame: Screening (Day-1) and Withdrawal (up to Study Week 129)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 269 | 265
Nanograms per milliliter (ng/mL)
  Screening, n=269, 265 | 58.6 (20.30) | 59.5 (44.20)
  Withdrawal, n=145, 157 | 59.0 (30.22) | 61.5 (16.74)

19. Secondary Outcome: Serum ErbB2 Concentration
Description: The Quest Laboratory collected blood samples for quantitative determination of serum ErbB2. The results of serum monitoring were used to compare tumor response rates following randomized therapy.
Time Frame: Screening (Day-1) and Withdrawal (up to Study Week 129)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 270 | 265
ng/mL
  Screening, n=270, 265 | 37.67 (95.883) | 36.19 (87.629)
  Withdrawal, n=145, 158 | 37.31 (98.257) | 39.95 (96.327)

20. Secondary Outcome: Number of Participants With the Indicated Adverse Events (AEs) With a Maximum Toxicity Grade of 3 or 4
Description: The severity of adverse events was graded per the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3. Grades 1 through 5 have unique clinical descriptions of severity for each AE based on the following general guideline: Grade 1, Mild AE; Grade 2, Moderate AE; Grade 3, Severe AE; Grade 4, Life-threatening or disabling AE; Grade 5, death related to AE.
Time Frame: Baseline (Day 1) until 30 days after the last dose of randomized therapy (average of 26 weeks)
Population: Safety Population: all randomized participants who received at least one dose of investigational product (based on the actual treatment received if this differed from that to which the participant was randomized). Two participants randomized to the placebo group actually received lapatinib.
Measure: Number; unit: participants
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Number analyzed (Participants) | 293 | 286
participants
  Diarrhea; Grade 3 | 43 | 4
  Diarrhea; Grade 4 | 1 | 0
  Alopecia; Grade 3 | 10 | 15
  Alopecia; Grade 4 | 0 | 0
  Rash; Grade 3 | 15 | 1
  Rash; Grade 4 | 0 | 0
  Nausea; Grade 3 | 7 | 2
  Nausea; Grade 4 | 0 | 0
  Myalgia; Grade 3 | 6 | 2
  Myalgia; Grade 4 | 0 | 0
  Neutropenia; Grade 3 | 30 | 20
  Neutropenia; Grade 4 | 23 | 14
  Vomiting; Grade 3 | 5 | 4
  Vomiting; Grade 4 | 0 | 0
  Arthralgia; Grade 3 | 7 | 4
  Arthralgia; Grade 4 | 0 | 0
  Fatigue; Grade 3 | 5 | 5
  Fatigue; Grade 4 | 0 | 0
  Asthenia; Grade 3 | 1 | 4
  Asthenia; Grade 4 | 1 | 0
  Neuropathy; Grade 3 | 7 | 3
  Neuropathy; Grade 4 | 0 | 0
  Decreased appetite; Grade 3 | 1 | 0
  Decreased appetite; Grade 4 | 0 | 0
  Pain in extremity; Grade 3 | 2 | 3
  Pain in extremity; Grade 4 | 2 | 0
  Peripheral sensory neuropathy; Grade 3 | 6 | 4
  Peripheral sensory neuropathy; Grade 4 | 0 | 0
  Pruritis; Grade 3 | 2 | 0
  Pruritis; Grade 4 | 0 | 0
  Paraesthesia; Grade 3 | 2 | 1
  Paraesthesia; Grade 4 | 0 | 0
  Constipation; Grade 3 | 0 | 0
  Constipation; Grade 4 | 0 | 0
  Cough; Grade 3 | 1 | 1
  Cough; Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and adverse events were collected from the first dose of randomized therapy until 30 days after the last dose of randomized therapy (average of 26 weeks).
Description: SAEs and AEs were collected in the Safety Population, comprised of all randomized participants who received at least one dose of investigational product (based on the actual treatment received if this differed from that to which the participant was randomized). Two participants randomized to the placebo group actually received lapatinib.
Arm/Group | Lapatinib With Paclitaxel | Placebo With Paclitaxel
Serious Adverse Events (participants affected / at risk) | 103/293 | 63/286
Other Adverse Events (participants affected / at risk) | 287/293 | 278/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib With Paclitaxel (N=293) | Placebo With Paclitaxel (N=286)
Neutropenia (Blood and lymphatic system disorders) | 22 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocythemia (Blood and lymphatic system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 24 | 2
Vomiting (Gastrointestinal disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischemia (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Device related infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 7 | 2
Mucosal inflammation (General disorders) | 6 | 1
Chest pain (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Edema peripheral (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 5 | 5
Hemoglobin decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Thrombosis (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Lumber radiculopathy (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib With Paclitaxel (N=293) | Placebo With Paclitaxel (N=286)
Alopecia (Skin and subcutaneous tissue disorders) | 153 | 183
Rash (Skin and subcutaneous tissue disorders) | 145 | 66
Pruritus (Skin and subcutaneous tissue disorders) | 46 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 5
Pain of skin (Skin and subcutaneous tissue disorders) | 4 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3
Rash generalized (Skin and subcutaneous tissue disorders) | 3 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 171 | 73
Nausea (Gastrointestinal disorders) | 100 | 85
Vomiting (Gastrointestinal disorders) | 74 | 48
Constipation (Gastrointestinal disorders) | 35 | 48
Dyspepsia (Gastrointestinal disorders) | 38 | 13
Abdominal pain (Gastrointestinal disorders) | 33 | 17
Stomatitis (Gastrointestinal disorders) | 21 | 13
Abdominal pain upper (Gastrointestinal disorders) | 12 | 16
Abdominal distension (Gastrointestinal disorders) | 14 | 9
Dry mouth (Gastrointestinal disorders) | 9 | 5
Hemorrhoids (Gastrointestinal disorders) | 6 | 4
Flatulence (Gastrointestinal disorders) | 5 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 5 | 2
Cheilitis (Gastrointestinal disorders) | 3 | 3
Epigastric discomfort (Gastrointestinal disorders) | 2 | 4
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 4 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Retching (Gastrointestinal disorders) | 1 | 3
Toothache (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1
Anal hemorrhage (Gastrointestinal disorders) | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0
Apthous stomatitis (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 1
Hematochezia (Gastrointestinal disorders) | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Diabetic gastropathy (Gastrointestinal disorders) | 1 | 0
Fecaloma (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal ischemia (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip edema (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 1
Melena (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Esophageal discomfort (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Parasthesia oral (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Tongue pigmentation (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 94 | 74
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 | 58
Pain in extremity (Musculoskeletal and connective tissue disorders) | 50 | 50
Bone pain (Musculoskeletal and connective tissue disorders) | 34 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 29
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 | 27
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 48 | 54
Paraesthesia (Nervous system disorders) | 43 | 42
Headache (Nervous system disorders) | 32 | 30
Neuropathy peripheral (Nervous system disorders) | 54 | 32
Dysgeusia (Nervous system disorders) | 12 | 11
Dizziness (Nervous system disorders) | 13 | 9
Hypoaesthesia (Nervous system disorders) | 11 | 10
Polyneuropathy (Nervous system disorders) | 9 | 3
Peripheral motor neuropathy (Nervous system disorders) | 8 | 4
Neuralgia (Nervous system disorders) | 3 | 4
Memory impairment (Nervous system disorders) | 3 | 3
Syncope (Nervous system disorders) | 3 | 2
Convulsion (Nervous system disorders) | 2 | 1
Neurotoxicity (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 2 | 0
Sinus headache (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0
Brain edema (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Coma hepatic (Nervous system disorders) | 0 | 1
Convulsions local (Nervous system disorders) | 0 | 1
Depressed level of consiousness (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neurophathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 65 | 61
Asthenia (General disorders) | 62 | 36
Pyrexia (General disorders) | 32 | 33
Mucosal inflammation (General disorders) | 38 | 9
Edema perpheral (General disorders) | 18 | 19
Pain (General disorders) | 19 | 16
Chest pain (General disorders) | 19 | 14
Chills (General disorders) | 6 | 8
Malaise (General disorders) | 6 | 7
Chest discomfort (General disorders) | 6 | 4
Axillary pain (General disorders) | 4 | 4
Influenza like illness (General disorders) | 4 | 5
Face edema (General disorders) | 4 | 2
Edema (General disorders) | 3 | 3
Catheter site pain (General disorders) | 1 | 2
Inflammation (General disorders) | 3 | 0
Adverse drug reaction (General disorders) | 0 | 2
Discomfort (General disorders) | 0 | 2
Injection site reaction (General disorders) | 1 | 1
Irritability (General disorders) | 0 | 2
Breakthrough pain (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 1 | 0
Catheter site related reaction (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Early satiety (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Implant site scar (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Infusion site edema (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Localized edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Vessel puncture site reaction (General disorders) | 1 | 0
Generalized edema (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 76 | 58
Anemia (Blood and lymphatic system disorders) | 32 | 35
Leukopenia (Blood and lymphatic system disorders) | 26 | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 4
Leukocytosis (Blood and lymphatic system disorders) | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Hyperchromasia (Blood and lymphatic system disorders) | 1 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 17 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 15
Urinary tract infection (Infections and infestations) | 15 | 8
Influenza (Infections and infestations) | 5 | 9
Pharyngitis (Infections and infestations) | 9 | 3
Cellulitis (Infections and infestations) | 4 | 5
Rhinitis (Infections and infestations) | 7 | 2
Pneumonia (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 5 | 4
Infection (Infections and infestations) | 6 | 1
Respiratory tract infection (Infections and infestations) | 5 | 2
Cystitis (Infections and infestations) | 2 | 4
Herpes simplex (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 3 | 3
Oral candidiasis (Infections and infestations) | 4 | 2
Device related infection (Infections and infestations) | 2 | 3
Folliculitis (Infections and infestations) | 3 | 2
Oral herpes (Infections and infestations) | 5 | 0
Acarodermatitis (Infections and infestations) | 4 | 0
Fungal infection (Infections and infestations) | 2 | 1
Laryngitis (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 1 | 3
Paronychia (Infections and infestations) | 5 | 0
Breast infection (Infections and infestations) | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Nail infection (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 2
Tonsillitis (Infections and infestations) | 3 | 0
Candidiasis (Infections and infestations) | 2 | 0
Catheter site infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Kidney infection (Infections and infestations) | 2 | 0
Lymphangitis (Infections and infestations) | 2 | 0
Otiits externa (Infections and infestations) | 2 | 0
Otitis media chronic (Infections and infestations) | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0
Breast abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Enterocolitis infection (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 3
Genital candidiasis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Omphalitis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 28
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 27 | 23
Aspartete aminotransferase increased (Investigations) | 22 | 20
Blood alkaline phosphatase increased (Investigations) | 19 | 19
Weight decreased (Investigations) | 17 | 14
Ejection fraction decreased (Investigations) | 6 | 6
Hemoglobin decreased (Investigations) | 8 | 4
Blood urea increased (Investigations) | 2 | 3
Weight increased (Investigations) | 1 | 9
Neutrophil count decreased (Investigations) | 5 | 3
White blood cell count decreased (Investigations) | 5 | 1
Body temperature increased (Investigations) | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 2
Blood albumin decreased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 2 | 2
Blood lactate dehydogenase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 2 | 1
Blood potassium decreased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 2
International normalized ratio increased (Investigations) | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood bilirubin decreased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood homocysteine increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood sodium increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Hemoglobin (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Prothrombin level decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 50 | 32
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 8
Dehydration (Metabolism and nutrition disorders) | 12 | 2
Hypokalemia (Metabolism and nutrition disorders) | 12 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 5 | 7
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperchloremia (Metabolism and nutrition disorders) | 0 | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1
Hyperproteinemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 34 | 29
Anxiety (Psychiatric disorders) | 13 | 13
Depression (Psychiatric disorders) | 10 | 13
Depressed mood (Psychiatric disorders) | 4 | 4
Confusional state (Psychiatric disorders) | 2 | 3
Restlessness (Psychiatric disorders) | 1 | 2
Hallucination (Psychiatric disorders) | 1 | 1
Mood altered (Psychiatric disorders) | 2 | 0
Eating disorder (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Personality disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Dysuria (Renal and urinary disorders) | 6 | 2
Hematuria (Renal and urinary disorders) | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Polyuria (Renal and urinary disorders) | 2 | 0
Enuresis (Renal and urinary disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 11 | 3
Drug hypersensitivity (Immune system disorders) | 3 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 6 | 4
Jaundice (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 7
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Immobile (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.